CLINICAL TRIAL: NCT05702437
Title: The Effects of Metabolic Syndrome and Its Components on Cognitive Performance and Physical Activity Level in Middle-age Individuals
Brief Title: Effect of MetS* on Cognitive Performance and Physical Activity (Metabolic Syndrome)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Aysenur Erekdag, Investigator, Istanbul University - Cerrahpasa
Other Study IDs: 3274238910
Record Dates: First submitted 2023-01-15; First posted 2023-01-27 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Metabolic Syndrome
Keywords: Cognitive Function; Physical Performance; Adults; Chronic Disease
MeSH Terms: conditions — Metabolic Syndrome; Chronic Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- MetS Group: it consists of volunteer participants diagnosed with MetS between the ages of 18 and 50. All assessments will be applied to the participants by two different researchers at the same time.
  Interventions: Other: assessment of cognitive performance
- Control Group: it will consist of healthy individuals aged 18-50 who do not have any health problems and have volunteered to participate in the study who have undergone a health check within the last 6 months.
  Interventions: Other: assessment of cognitive performance

INTERVENTIONS:
Other: assessment of cognitive performance — evaluation of the cognitive and physical performance of the participants by two separate researchers at the same time
  Other Names: assessment of physical performance

SUMMARY:
Metabolic syndrome (MetS) increases the risk of developing diabetes and cardiovascular disease risk factors that are linked with each other, which is a metabolic dysfunction, which contains a combination of multiple.

It is known that METS plays a role in the development of many diseases such as cardiovascular diseases, stroke, cancer, Alzheimer's. Studies have revealed that neuroinflammation, oxidative stress, abnormal lipid metabolism and impaired vascularization, which play a role in the pathogenesis of MetS, affect the structure of the brain and cognition. Atherosclerosis of the carotid artery, increased brain atrophy and white matter damage are potential explanatory mechanisms that lead to an impact on cognitive skills in patients with MetS. In addition, the existence of MetS components such as obesity, diabetes, hypertension alone also negatively affects cognitive functions, and the level of cognitive influence also increases as the number of components an individual has increases.

The literature reports that learning, executive functions, processing speed, attention/working memory and global cognitive functions are affected in individuals with MetS, but no consensus has been reached on this issue. Some studies say that MetS causes a significant decrease in cognitive functions, while some studies indicate that this difference is not significant.

The aim of our study is to proof the relationship between MetS and cognitive functions with metabolic syndrome components.

H1:There is a relationship between the MetS and cognitive functions.

DETAILED DESCRIPTION:
Voluntary participants who have been diagnosed with MetS and agreed to voluntary health subjects will be included in the study. Signed voluntary consent will be obtained from participants. Participants will be divided into two groups. There will be individuals diagnosed with MetS in the intervention group and healthy individuals who do not have any problems in the control group.

ELIGIBILITY:
Inclusion Criteria:

* being between the ages of 18-50
* Having been educated for at least 5 years and know how to read and write
* Having been diagnosed with MetS by meeting 3 of the NCEP-ATP III criteria (for participants in the MetS Group)
* To have a biochemistry test performed within the last 6 months (for the Healthy Group)
* Not having any MetS components (For the Healthy Group)

Exclusion Criteria:

* Having any neurological, psychiatric and psychological diseases that may affect cognitive status
* Taking antipsychiatric medication
* The presence of any visual-auditory intellectual disability
* Having undergone bariatric surgery

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Men and women who have been diagnosed with MetS according to NCEP-ATP III criteria and healthy individuals who do not have any health problems
Sampling Method: Probability Sample
Enrollment: 82 (Estimated)
Dates: Start 2023-02-20 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Evaluation of Metabolic Syndrome-waist circumference | once, at baseline
  Waist Circumference measurement will be recorded with a tape measure in the middle between the last palpable rib and the upper edge of the iliac crest.
Evaluation of Metabolic Syndrome-blood pressure | once, at baseline
  "Omron" digital blood pressure monitor will be used to measure systolic and diastolic blood pressure. Participants will be asked to rest for 5 minutes before the measurement.
Evaluation of Metabolic Syndrome-triglyceride | once, at baseline
  Triglyceride, HDL-C and fasting plasma levels and biochemistry laboratory findings of individuals will be evaluated. Before the analysis, 8-12 hours of fasting is required so that it does not affect the test results.
Evaluation of Metabolic Syndrome-HDL-C | once, at baseline
  Triglyceride, HDL-C and fasting plasma levels and biochemistry laboratory findings of individuals will be evaluated. Before the analysis, 8-12 hours of fasting is required so that it does not affect the test results.
Evaluation of Metabolic Syndrome-fasting plasma level | once, at baseline
  Triglyceride, HDL-C and fasting plasma levels and biochemistry laboratory findings of individuals will be evaluated. Before the analysis, 8-12 hours of fasting is required so that it does not affect the test results.
Metabolic Syndrome Severity Score | once, at baseline
  This scoring creates a z-score by considering factors such as age, race, gender, and metabolic syndrome components values. There is a website that automatically calculates the z-score when these data are entered. (https://metscalc.org/metscalc/)
Monreal Cognitive Assessment | once, at baseline
  This scale consists of parts that evaluate executive functions, attention and concentration, memory, language, abstract thinking, visual-spatial skills, orientation and calculation. The application of MoCA takes about 10 minutes and the total score of the scale is calculated over 30 points. The threshold point value is 21. Scores of 20 or less are considered cognitive dysfunction.
Stroop Test TBAG Form | once, at baseline
  a neuropsychological test that measures focused attention and the speed of information processing

SECONDARY OUTCOMES:
Mini Mental State Examination | once, at baseline
  it is a test consisting of 11 questions that evaluate different cognitive parameters, including recording memory, attention and calculation, recall and language, motor function and perception. The maximum score that can be taken from the test is 30 and there is no time limit. In scoring, 24-30 points are normal, 23 points and below indicate mild cognitive impairment.
Visual Reaction Test | once, at baseline
  the participant sees a red circle appearing on a white screen on the computer at variable time intervals and should press the December key of the computer quickly as soon as he sees the circle.
International Physical Activity Questionnare Short-Form | once, at baseline
  taking into account the last week, the time spent on walking, moderate and vigorous activities is questioned.
pedometer | once, at baseline
  A valid and reliable method for comparing the participants' weekly step counts and determining their physical activity levels

CONTACTS AND LOCATIONS:
Overall Officials: Ayca Arslanturk, BSc, Principal Investigator — Bezmialem Vakif University
Locations (1):
- Bezmialem Vakif University, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Fahed G, Aoun L, Bou Zerdan M, Allam S, Bou Zerdan M, Bouferraa Y, Assi HI. Metabolic Syndrome: Updates on Pathophysiology and Management in 2021. Int J Mol Sci. 2022 Jan 12;23(2):786. doi: 10.3390/ijms23020786. PMID 35054972
- [Background] Expert Panel on Detection, Evaluation, and Treatment of High Blood Cholesterol in Adults. Executive Summary of The Third Report of The National Cholesterol Education Program (NCEP) Expert Panel on Detection, Evaluation, And Treatment of High Blood Cholesterol In Adults (Adult Treatment Panel III). JAMA. 2001 May 16;285(19):2486-97. doi: 10.1001/jama.285.19.2486. No abstract available. PMID 11368702
- [Background] Bahchevanov KM, Dzhambov AM, Chompalov KA, Massaldjieva RI, Atanassova PA, Mitkov MD. Contribution of Components of Metabolic Syndrome to Cognitive Performance in Middle-Aged Adults. Arch Clin Neuropsychol. 2021 May 21;36(4):498-506. doi: 10.1093/arclin/acaa081. PMID 33067992
- [Background] Tahmi M, Palta P, Luchsinger JA. Metabolic Syndrome and Cognitive Function. Curr Cardiol Rep. 2021 Oct 19;23(12):180. doi: 10.1007/s11886-021-01615-y. PMID 34668083
- [Background] Wichayanrat W, Boripuntakul S, Keawtep P, Worakul P, Sungkarat S. Obesity and Brain Health: The Impact of Metabolic Syndrome and Cardiorespiratory Fitness on Cognitive Performances in Middle-Aged Obese Women. J Prev Alzheimers Dis. 2022;9(4):701-707. doi: 10.14283/jpad.2022.54. PMID 36281674